CLINICAL TRIAL: NCT04257409
Title: Musculoskeletal Changes Induced by Physiotherapeutic Intervention, and Their Impact on the Induction of Diabetic Foot Syndrome and Psychosocial Status in Type 2 Diabetes Mellitus
Brief Title: Musculoskeletal Changes After Physiotherapeutic Intervention in Podiatric Subjects
Acronym: BIONEDIAN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mgr. Eliška Vrátná (Other)
Collaborators: Vladimíra Fejfarová, MD, PhD (Unknown); prof. Ing. Václav Bunc, CSc (Unknown)
Responsible Party: Sponsor-Investigator, Mgr. Eliška Vrátná, Faculty of Physical Education and Sport, Charles University, Czech Republic
Organization: Charles University, Czech Republic (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 546417
Record Dates: First submitted 2019-12-15; First posted 2020-02-06 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Prevention of Diabetic Foot
Keywords: diabetic foot; biomechanics; quality of life; prevention
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: 60 patients with Type 2 diabetes mellitus. These patients will be randomized into 3 study groups - patients with type 2 DM with mild form of peripheral sensory neuropathy (20 subjects), patient with severe peripheral neuropathy (20 subjects) and those with diabetic foot syndrome, without active lesion (20 subjects). All patients will undergo 12 week lasting active intervention program consisting of recommendations by a physiotherapist focusing on the improvement of physical fitness, muscle strength and foot joint improvement. Control group will be consisted of 20 patients with healed diabetic foot.
Who Masked: Participant
Masking Description: randomization of diabetic patients with healed diabetic foot according the randomization scheme
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- DF patient active (Experimental): Patients with Type 2 diabetes mellitus and diabetic foot, whose have healed diabetic foot ulcers
  Interventions: Other: Physical intervention by exercise
- DF patient control (Active Comparator): Patients with Type 2 diabetes mellitus and diabetic foot, whose have healed diabetic foot ulcers
  Interventions: Other: Physical intervention by exercise
- Diabetic patient with mild neuropathy (Experimental): Patients with Type 2 diabetes mellitus with mild form of peripheral sensory neuropathy
  Interventions: Other: Physical intervention by exercise
- Diabetic patient with severe neuropathy (Experimental): Patients with Type 2 diabetes mellitus with severe form of peripheral sensory neuropathy
  Interventions: Other: Physical intervention by exercise

INTERVENTIONS:
Other: Physical intervention by exercise — 12 week lasting exercise intervention

SUMMARY:
The recurrence of diabetic foot ulcers (DFU) is a key problem in podiatric care. It is very often given by biomechanical abnormalities frequently present in those patients. The aim of our randomized controlled study is to find possible changes as of plantar pressures as of biomechanics of the ankle and small joints in patients with type 2 diabetes mellitus with different degrees of neuropathy. During this project, investigators will examine the possible impact of 12-week lasting intervention program on the distribution of plantar pressures, joint mobility and muscle strength of lower limbs. The incidence of ulcerations / reulcerations and changes of psychosocial characteristics will be evaluated during the study period.

Approximately 60 patients with Type 2 diabetes mellitus will be included into the study. These patients will be randomized into 3 study groups - patients with type 2 DM with mild form of peripheral sensory neuropathy (20 subjects), patient with severe peripheral neuropathy (20 subjects) and those with diabetic foot syndrome, without active lesion (20 subjects). All patients will undergo 12 week lasting active intervention program consisting of recommendations by a physiotherapist focusing on the improvement of physical fitness, muscle strength and foot joint improvement. Control group will be consisted of 20 patients with healed diabetic foot.

The outcomes of this project will try to objectively verify in the randomized controlled trial the impact of exercise on lower limb biomechanics, mobility, self-sufficiency, quality of life in patients with type 2 diabetes mellitus at risk or already developed diabetic foot syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* sensoric neuropathy (mild - based on VPV 15-30 V or EMG results, severe - based on VPT above 50 V or EMG results)
* diabetic foot with healed diabetic foot ulcers, inactive Charcot foot

Exclusion Criteria:

* impossibility to exercise
* amaurosis
* non-compliance
* critical limb ischemia
* active ulcer, surgical wound
* active Charcot foot
* active carcinoma
* recent stroke (last 8 weeks)
* recent myocardial infarction (last 8 weeks)
* recent PTA, PCI, bypass (last 8 weeks)
* myopathy
* rheumatoid arthritis
* cox-, gonartrosis of 3rd -4th grade.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 30-75 years
Enrollment: 80 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-03-30 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Biomechanics- plantar pressures | changes after 12 weeks, 24 weeks
  plantar pressures will be evaluated by pedobarograph (in Newtons)
Biomechanics- biomechanics of the ankle | changes after 12 weeks, 24 weeks
  biomechanics of the ankle will be assessed by goniometry in angles
Biomechanics- changes of foot joint angles | changes after 12 weeks, 24 weeks
  changes of foot joint agles will be evaluated by measurement of X-Rays bones angles - calcaneal pitch, talar-1st metatarsal angle and lateral Talocalcaneal angle
Fitness - physical activity | changes after 12 weeks, 24 weeks
  The amount of physical activity will be assessed by IPAQ questioners
Fitness - muscle strength | changes after 12 weeks, 24 weeks
  Muscle strength will be measured by dynamometry in Newtons
Fitness - senior fitness | changes after 12 weeks, 24 weeks
  fitness will be assessed by seniorfittest containing 2 minutes step test (steps/2 min) and test of sitting (sits/30 seconds)

SECONDARY OUTCOMES:
ulceration/reulceration | changes after 12 weeks, 24 weeks
  detection of the incidence of ulceration/reulceration
Psychosocial changes - quality of life | changes after 12 weeks, 24 weeks
  Quality of life will be evaluated by WHO-QoL Bref test (4 domains - high values mean bettr findings
Psychosocial changes - depression | changes after 12 weeks, 24 weeks
  Depression status will be asessed by Geriatric Depression Scale (GDS) scale - minimum 0, maximum 30 points (higher then 9 points- mild form of depression, higher then 20 - severe depression
Psychosocial changes - stress readaptation | changes after 12 weeks, 24 weeks
  Adaptation to stress will be detected by Stress Readaption Scale (0-400 points) - points higher then 150 - higher risk of worse stress readaptation and therefore higher risk of somatisation
Metabolism - glucose control | changes after 12 weeks, 24 weeks
  Investigators will be loked for metabolic changes in diabetes control (HbA1c in mmol/mol, glycemia in mmol/l)
Metabolism - lipid profile | changes after 12 weeks, 24 weeks
  The authors will control lipid profiles (Total-, HDL-, LDL-cholesterol in umol/l)
Metabolism - myokines | changes after 12 weeks, 24 weeks
  Patients will be checked for changes in selected cytokines nad myokines (IL-4,6,7,8,15 in pg/ml, myostatin in pg/ml, irisin in ng/ml, FGF-21 in pg/ml)

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Clinical and Experimental Medicine, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Undecided
Possible to look at the data in documentation site